CLINICAL TRIAL: NCT01900158
Title: A Phase I/II Dose Escalation Study to Assess the Safety, Tolerability and Efficacy of Amphinex®-Induced Photochemical Internalisation (PCI) of Gemcitabine in Patients With Advanced Inoperable Cholangiocarcinomas
Brief Title: A Phase I/II Safety and Efficacy Study of PCI of Gemcitabine and Chemotherapy in Patients With Cholangiocarcinomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PCI Biotech AS (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PCI A202/12; 2012-002888-10 (EudraCT Number)
Record Dates: First submitted 2013-05-15; First posted 2013-07-16 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2019-08

CONDITIONS: Cholangiocarcinoma
Keywords: Phase I; CCA; Cholangiocarcinoma; bile duct cancer; klatskin; perihilar; Amphinex; Gemcitabine; Photochemical internalisation; Safety; Tolerability; Efficacy; Cisplatin; PCI; extrahepatic; local control; local tumour treatment; biliary; fimaporfin
MeSH Terms: conditions — Cholangiocarcinoma; Bile Duct Neoplasms | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Intervention Model Description: Phase I Dose escalation study With 4 cohorts of different doses of light and fimaporfin (Dose Escalation) plus and additional cohort With one repeated treatment of the dose selected for one treatment (Extended).
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase I (Experimental): Experimental PCI treatment in dose escalation cohorts consist of Amphinex injection (at different doses) plus a single standard dose of Gemcitabine (1000 mg/m2) plus intraluminal light at the tumour area (at different doses). In addition up to 8 cycles of standard chemotherapy doses of Gemcitabine (1000 mg/m2) and Cisplatin (25 mg/m2) was provided. In the Extended part of the study (last cohort) an additional PCI treatment was introduced at Cycle 5 in the treatment Schedule.
  Interventions: Drug: Amphinex, Gemcitabine and Cisplatin

INTERVENTIONS:
Drug: Amphinex, Gemcitabine and Cisplatin — Amphinex administration on day 0, followed by gemcitabine administration (1000 mg/m2) and laser light application (652 nm) on day 4 followed by systemic gemcitabine (1000 mg/m2) and cisplatin (25 mg/m2) given on Day 1 and Day 8 of each 21-day cycle, for up to a total of eight cycles. Either one or two PCI treatments (Amphinex, Gemcitabine and intraluminal laser light of 652nm) during the 8 cycles of chemotherapy
  Other Names: Gemzar (Gemcitabine); Fimaporfin (Amphinex); Cisplatin

SUMMARY:
This is a Phase I Dose Escalation Study in which the safety, tolerability and efficacy of Amphinex®--induced Photochemical Internalisation (PCI) of Gemcitabine followed by Gemcitabine/Cisplatin Chemotherapy will be assessed in patients with advanced inoperable cholangiocarcinomas.

DETAILED DESCRIPTION:
Cholangiocarcinoma (CCA) is an uncommon adenocarcinoma arising from the neoplastic transformation of cholangiocytes, the epithelial cells lining the intra-hepatic and extra-hepatic bile ducts. CCA accounts for about 3% of all digestive tumours and 10-15% of the hepatobiliary tumours. It has an annual incidence of 1-2 cases per 100,000 in the Western World, but rates of CCA have been steadily rising worldwide over the past several decades. On a global scale, CCA is the second most common primary hepatic malignancy These tumours have a poor overall survival with a 5-year survival of about 5%. Over 50% of patients present with advanced-stage disease, and the prognosis is poor with the survival of between 6-12 months for unresected patients, even after biliary decompression. CCA may arise anywhere in the biliary tree, from the small, peripheral hepatic ducts to the distal common bile duct. Commonly used classification systems utilise anatomical location to group tumours into three main categories: intra-hepatic (20-25%), perihilar (also including hilar/Klatskin tumour - 50%) and distal (20-25%).

Hilar CCA is an adenocarcinoma of the extrahepatic biliary tree arising from the main left or right hepatic ducts or their confluence. There has a been a growing recognition that hilar CCA disease actually has a distinct biological behaviour and natural history compared to that of (distal) extra-hepatic CCA, and increasing acknowledgment that different therapeutic strategies are required. At initial presentation of patients with extra-hepatic CCA, 30-50% will have local lymph node involvement and 10-20% metastatic spread typically to the liver and peritoneum. With hilar CCA due to the long asymptomatic course, only 20% are resectable at time of diagnosis.

Standard treatment options for CCA include surgery, radiotherapy and chemotherapy, dependent upon if the CCA is intra- or extra-hepatic. Tumour resection is the only potential cure for CCA. Recent advances in transplantation using stringent selection criteria and utilization of neoadjuvant chemoradiation have demonstrated encouraging results with 5 year survival rates of over 70%, with even one series from The Mayo Clinic yielding a 5-year survival rate of 82%. For the 80% who present with unresectable disease, the utility of these modalities combined with biliary decompression interventions only provided a median survival time of 3-6 months from the time of diagnosis.

For these patients with inoperable advanced CCA the main treatment aim is palliative to relieve local symptoms such as pain and jaundice. Surgery for these patients is primarily for creating a bypass in patients who cannot be stented. CCA is remarkably resistant to pharmacological therapy, but activity has been seen using chemotherapy; mainly gemcitabine given either as monotherapy or paired with either a platin derivative or a fluoropyrimidine as a doublet treatment and more recently docetaxel, these give partial response (PR) rates of 0-9% and an average survival advantage of 2-12 months. Concerning biological therapy, the ongoing studies using sorafenib, lapatinib or bevacizumab have yielded some promising results, with sorafenib demonstrating therapeutic benefit in a single arm Phase II study. For patients who are unsuitable for curative resection, the current systemic combination chemotherapy is with cisplatin plus gemcitabine. This was established in the largest randomized phase III study to date in non-operable biliary tract cancer which demonstrated a response rate of 81.4% and a median overall survival (OS) of 11.7 months; notably there was no statistically significant increase in toxicity when compared to gemcitabine monotherapy. The recent advances in interventional and endoscopic technology have seen a rise in highly specialized centres that are able to deliver very precise local control treatments aimed at gaining local control; these include local ablation and embolization, brachytherapy, radio-frequency ablation and, most significantly, photodynamic therapy which (PDT), with its favourable adverse-event profile, is recommended by most recent review articles for non-resectable patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically/cytologically (C5) verified adenocarcinoma consistent with cholangiocarcinoma
2. Cholangiocarcinoma that:

   * Is considered to be inoperable
   * Has a primary lesion in the perihilar biliary duct region that requires stent placement
   * Has nodal enlargement ≤ to N1 as per CT/MRI assessment
   * If has metastatic disease; this should be confined to the liver parenchyma only
3. Adequate biliary drainage (either at least 50% of the liver volume, or at least two sectors), with no evidence of active uncontrolled infection (patients on antibiotics are eligible).
4. Age ≥ 18 years.
5. Performance status ECOG ≤ 1.
6. Estimated life expectancy of at least 12 weeks.
7. Written informed consent.

Exclusion Criteria:

1. Any prior anti-cancer (either local or systemic) treatment for cholangiocarcinoma.
2. Patients with extra-hepatic metastatic cholangiocarcinoma.
3. Patients with a severe visceral disease other than cholangiocarcinoma.
4. Patients with primary sclerosing cholangitis.
5. Patients with porphyria or hypersensibility to porphyrins.
6. Patients with an active second primary cancer, with exception of adequately treated basal cell carcinoma, squamous cell carcinoma or other non-melanomatous skin cancer, or in-situ carcinoma of the uterine cervix. An active second primary cancer is defined as one with a disease-free interval of < 5 years before registration/randomization.
7. Inability to undergo CT or MRI.
8. Current participation in any other interventional clinical trial.
9. Male patients not willing to use adequate contraception or female patients of childbearing potential not willing to use an effective form of contraception such as hormonal birth control, intrauterine device or double barrier method during PCI treatment and subsequent chemotherapy and for at least 6 months thereafter.
10. Breast feeding women or women with a positive pregnancy test at baseline.
11. Inadequate bone marrow function:

    Absolute Neutrophil Count (ANC): < 1.5 x 10^9/L, or platelet count < 100 x 10^9/L or haemoglobin < 6 mmol/L (transfusion allowed).
12. Inadequate liver function, defined as:

    * Serum (total) bilirubin > 2.5 x the Upper Limit of Normal (ULN) for the institution.
    * Aspartate Amino Transferase (AST) or Alanine Amino Transferase (ALT) > 3.0 x ULN (> 5 x ULN if liver metastases are present)
    * Alkaline phosphatase (ALP) levels > 5.0 x ULN.
13. Inadequate renal function, defined as:

    Creatinine clearance < 60 mL/min
14. Planned surgery, endoscopic examination or dental treatment in the first 30 days after PCI treatment.
15. Co-existing ophthalmic disease likely to require slit-lamp examination within the first 90 days after PCI treatment.
16. Clinically significant and uncontrolled cardiac disease including unstable angina, acute myocardial infarction within six months prior to baseline, congestive heart failure, and arrhythmia requiring therapy, with the exception of extra systoles or minor conduction abnormalities and controlled and well treated chronic atrial fibrillation.
17. Known allergy or sensitivity to photosensitisers.
18. Ataxia telangiectasia.
19. Evidence of any other medical conditions (such as psychiatric illness, infectious diseases, physical examination or laboratory findings) that may interfere with the planned PCI treatment, affect patient compliance or place the patient at high risk from treatment-related complications.
20. Significant hearing impairment.
21. Patients concurrently receiving phenytoin.
22. Patients defined as vulnerable according to French law (France only)
23. Patients using or have been using photosensitising drugs within the last 7 days (France only)
24. Patients who have received amiodarone in the last year (France only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLT) and the safety profile | up to 6 months
  Clinically significant toxicity or abnormal laboratory value assessed as unrelated to the underlying disease, criteria's based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.02:
  * Photosensitivity Grade 3 outside the treatment area, except for areas exposed for skin sensitivity tests and areas exposed for re-introduction to normal light. Patient compliance with light protection guidelines MUST be followed; noncompliance will be taken into account
  * Phototoxicity Grade 4 inside the treatment area (e.g., duodenal ulceration).
  * Non-haematological toxicity (excluding nausea and vomiting) ≥Grade 3.
  * Neutropenia or thrombocytopenia Grade 4.
  * All other Grade 3 toxicities that are clinically unexpected.
Schedule-limiting toxicities (SLTs) and the safety profile | up to 6 months
  Clinically significant toxicity or abnormal laboratory value assessed as unrelated to the underlying disease criteria's based on the NCI CTCAE version 4.02:
  * Photosensitivity Grade 3 outside the treatment area, except for areas exposed for skin sensitivity tests and areas exposed for re-introduction to normal light despite following prescribed precautions. Patient compliance with light protection guidelines MUST be followed; noncompliance will be taken into account
  * Clinically significant phototoxicity inside the treatment area (e.g., duodenal ulceration, cholangitis or pancreatitis requiring interventional radiology, operative intervention or would lead to such intervention including events that would have life-threatening consequences)
  * A toxicity of any grade that is clinically unexpected and considered related to the PCI treatment (changes to cisplatin treatment alone will not be included as part of this assessment).

SECONDARY OUTCOMES:
Measuring the Amphinex and Gemcitabine concentration in blood plasma | Up to 8 months
  Cmax, Vss, T1/2, AUC and CL
Progression-free survival (according to RECIST 1.1 criteria) | Up to documented disease progression or death (or Database lock)
Best Overall Response (according to RECIST 1.1 criteria) | Up to Database lock

OTHER OUTCOMES:
Time to re-intervention (stent patency) | Up to 8 months
  From date of registration to reintervention
Patient questionnaire and "in clinic" evaluations | Up to 8 months
  Skin photosensitivity - protection information- testing information and events
Measuring of Amphinex concentration in faeces | up to 1 week after Amphinex administration
  Quantitative measures
Local tumor response evaluation | Up to 8 months
  Local tumour responses by assessment of radiological data

CONTACTS AND LOCATIONS:
Overall Officials: Dr Richard Sturgess, MD, Principal Investigator — University Hospital Aintree
Locations (11):
- CHU Angers, Angers, Maine-et-Loire, France
- Germany (8):
  - Klinikum rechts der Isar, Technische Universität München, Munich, Bavaria
  - Klinikum der Ludwig-Maximilians-Universität, München, Bavaria
  - Klinikum der Johann Wolfgang Goethe-Universität, Frankfurt am Main, Hesse
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Klinikum Ludwigshafen, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Charité, Campus Mitte, Berlin
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden
- Oslo Universtiy Hospital, Oslo, Norway
- University Hospital Aintree, Aintree, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor — http://www.pcibiotech.no